CLINICAL TRIAL: NCT05278975
Title: A Translational Phase 1/2 Dose-Escalation and Expansion Study to Determine Safety, Tolerability, and Recommended Phase 2 Dose of RSO-021 in Patients With Malignant Pleural Effusion Due to Advanced/Metastatic Solid Tumors Including Mesothelioma
Brief Title: Study of RSO-021 in Patients With Malignant Pleural Effusion Due to Advanced/Metastatic Solid Tumors Including Mesothelioma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RS Oncology LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RS-TS-101-01
Record Dates: First submitted 2022-02-07; First posted 2022-03-15 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Malignant Pleural Effusion; Malignant Pleural Mesothelioma; Mesothelioma; Mesotheliomas Pleural; Mesothelioma; Lung; Pleural Effusion, Malignant
MeSH Terms: conditions — Pleural Effusion, Malignant; Mesothelioma, Malignant; Mesothelioma | interventions — Thiostrepton

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Phase 1 - Dose Escalation (Experimental): RSO-021 administered in increasing doses as a solution for pleural infusion through an indwelling IP catheter, administered as a single dose on Day 1 of each week of a 21-day treatment cycle.
  Interventions: Drug: RSO-021
- Ph2 - Dose Expansion - MPE from non-mesothelioma solid tumors (Experimental): RSO-021 administered at the MTD/RP2D as a solution for pleural infusion through an indwelling IP catheter, administered as a single dose on Day 1 of each week of a 21-day treatment cycle in patients with MPE from non-mesothelioma solid tumors.
  Interventions: Drug: RSO-021
- Ph2 - Dose Expansion - MPE from mesothelioma (Experimental): RSO-021 administered at the MTD/RP2D as a solution for pleural infusion through an indwelling IP catheter, administered as a single dose on Day 1 of each week of a 21-day treatment cycle in patients with MPE from mesothelioma.
  Interventions: Drug: RSO-021
- P2 - Dose Expansion - mesothelioma -First line treatment prior to Ipi/Nivo (Experimental): RSO-021 administered at the MTD/RP2D as a solution for pleural infusion through an indwelling IP catheter, administered as a single dose on Day 1 of each week of a 21-day treatment cycle in patients with mesothelioma. This local treatment with RSO-021 is prior to systemic treatment of Ipi/Nivo.
  Interventions: Drug: RSO-021
- Ph2 - Dose Expansion - MPE from non-mesothelioma solid tumors combination with Paclitaxel (Experimental): RSO-021 administered at the MTD/RP2D as a solution for pleural infusion through an indwelling IP catheter, administered as a single dose on Day 1 of each week of a 21-day treatment cycle in patients with MPE from non-mesothelioma solid tumors. In combination with Paclitaxel. Paclitaxel will be administered as a systemic therapy per SoC and the approved labeling based on the tumor type being treated. Paclitaxel is commercially available in the UK
  Interventions: Drug: RSO-021

INTERVENTIONS:
Drug: RSO-021 — A naturally-occurring, sulfur-rich, cyclic oligopeptide antibiotic of the thiopeptide class.
  Other Names: Thiostrepton

SUMMARY:
This is an open-label, non-randomized, multicenter, translational Phase 1/2 dose-escalation and expansion study designed to determine the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary anti-tumor activity of RSO-021 after intrapleural (IP) administration in patients with malignant pleural effusion (MPE) (non-mesothelioma) and MPE from mesothelioma.

DETAILED DESCRIPTION:
This is a Phase 1/2, open-label, multi-center study whose primary Phase 1 stage objective is to determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of RSO-021 (thiostrepton), a naturally-occurring, sulfur-rich, cyclic oligopeptide antibiotic of the thiopeptide class, in patients with MPE from any solid tumor, including mesothelioma.

In the Phase 2 stage, once the RP2D has been identified, the antitumor activity of RSO-021 will be evaluated in four recruitment arms; (1) in patients with MPE (non-mesothelioma), (2) in patients with MPE (non-mesothelioma) in combination with paclitaxel, (3) in patients with MPE from mesothelioma after first-line SoC, and (4) in patients with MPE from mesothelioma who have a 'window of opportunity' for treatment prior to first-line systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years old.
2. ECOG performance status 0-1.
3. Histological diagnosis of solid tumor/mesothelioma with MPE.

   Expansion Cohort 2:
   1. only patients with breast cancer, ovarian cancer or non-small cell lung cancer.
   2. patients for whom paclitaxel is a recommended SoC therapy.
   3. no contraindications to paclitaxel.
4. Patients with a disease burden that is predominantly pleural, and a pleural space that is accessible.

Expansion Cohorts 1 and 2: MPE (non-mesothelioma): patients must have received at least 1 prior standard of care treatment regimen for advanced, unresectable malignancy, with documented progression.

Expansion Cohort 3:

MPE mesothelioma: patients must have received at least 1 prior standard-of-care treatment regimen for advanced, unresectable malignancy, with documented progression and there is no approved life extending alternative available.

Expansion Cohort 4: MPE mesothelioma 'window of opportunity': patients should be treatment naïve, have refused or not be immediately requiring of systemic therapy and should be patients for whom drainage is planned immediately while further treatment options are arranged. It must be documented for each patient that protocol participation will not affect their subsequent ability to access standard systemic first line therapy due to RSO-021 being a local therapy.

6. Resolution of all acute reversible toxic effects of prior therapy or surgical procedure to Grade ≤1 (except alopecia).

7. For dose escalation: Archival paraffin block, ideally from the patient's most recent biopsy, should be provided prior to the first dose of study therapy, if sufficient tissue is available.

For dose expansion cohorts: fresh tumor biopsy must be obtained.

1. Patients enrolled in the mesothelioma expansion phase will be requested to undergo a tumor biopsy during the screening period and after the third dose.
2. Patients enrolled in the non-mesothelioma expansion phase will be requested to undergo a tumor biopsy during the screening period and after the third dose only if medically feasible.

   8. Patients must have adequate organ function.

Exclusion Criteria:

1. Last dose of prior anti-cancer therapies:

   1. Systemic anti-cancer therapy within 3 weeks or 5 half-lives prior to study entry, whichever is shorter.
   2. Thoracic radiation therapy or significant surgery within 3 weeks prior to study entry. Localized palliative radiotherapy for pain control in non-target lesions is allowed during the screening period.
   3. Received an investigational product or been treated with an investigational device within 30 days prior to first drug administration or plans to participate in any other clinical trial while on this study.
2. Previous or concurrent malignancy that would prevent evaluation of the primary endpoint (e.g. R/R hematological malignancy).
3. Patients whose extent of tumor or loculations would render intrapleural administration incomplete and/or ineffective.
4. Known hypersensitivity to the active ingredient or any excipient contained in the drug formulation.
5. History or clinical evidence of any surgical or medical condition which the investigator and/or medical monitor judges as likely to interfere with the results of the study or pose an additional risk in participating, e.g., rapidly progressive or uncontrolled disease involving a major organ system-vascular, cardiac, pulmonary, gastrointestinal, gynecologic, hematologic, neurologic, neoplastic, renal, endocrine, or an immunodeficiency, or clinically significant active psychiatric or abuse disorders.
6. Active infection with human immunodeficiency virus (HIV) and CD4+ T-cell count < 350/μL. Patients not on established anti-retroviral therapy for at least four weeks prior to first dose of study drug and having a detectable HIV viral load. Testing is not required for eligibility.
7. Active infection with hepatitis B (surface antigen); or infection with hepatitis C in absence of sustained virologic response. Testing is not required for eligibility.
8. Pregnant or breast-feeding patients.
9. Patients with symptomatic or unstable CNS primary tumor or metastases and/or carcinomatous meningitis. Patients with documented treated CNS metastases stable off steroids may be enrolled at the discretion of the investigator.
10. Therapeutic oral anticoagulation for a thromboembolic event (prophylactic anticoagulation is allowed as long as patient can undergo catheter placement and biopsy). LMWH is allowed on condition that it is medically acceptable to interrupt LMWH therapy for all study procedures.
11. Use of systemic corticosteroids to treat inflammatory or autoimmune symptoms within 15 days or other immunosuppressive drugs within 3 weeks prior to start of the study. Inhaled and topical corticosteroids are permitted. Up to 10 mg/day prednisone or equivalent is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicity | First 21 days of treatment.
  The incidence of DLTs during the DLT assessment period.
Frequency and Severity of Adverse Events (AE) | Screening to 90 days from last dose.
  The incidences and percentages of patients experiencing AEs summarized by NCI CTCAE version 5.0 grade and by causality.
Dose Finding | Screening to 90 days from last dose.
  Determination of the MTD and/or the RP2D.

SECONDARY OUTCOMES:
Pharmacokinetics of RSO-021 | Day 1 of dosing through 21 days post last dose.
  Maximum Plasma Concentration (Cmax)
Pharmacokinetics of RSO-021 | Day 1 of dosing through 21 days post last dose.
  Area Under the Curve (AUC)
Objective Response Rate (ORR) | Day 1 of dosing through day 90 after the last dose.
  ORR according to RECIST v1.1.
Disease Control Rate (DCR) | Day 1 of dosing through day 90 after the last dose.
  The percentage of subjects with a complete response, partial response, or stable disease for at least 2 consecutive tumor assessments.
Progression Free Survival (PFS) | Day 1 of dosing through day 90 after the last dose.
  Time from the date of initiation of study therapy to the date measurement criteria are first met for PD or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: James Spicer, MD, Principal Investigator — Guys Hospital
Locations (10):
- United Kingdom (10):
  - South Mead North Bristol Hopsital, Bristol
  - NHS Greater Glasgow & Clyde, Glasgow
  - Leeds Teaching Hospital, Leeds
  - Facility: HOPE Clinical Trials Facility, Leicester Royal Infirmary, Leicester
  - Barts Health NHS Cancer Institute, London
  - Guys and St Thomas NHS Foundation Trust, London
  - The Royal Marsden, London
  - The Christie NHS, Manchester
  - Northumbria NorthTyne Side General Hospital, North Shields
  - Oxford University Hospitals NHS Foundation, Oxford

IPD SHARING:
Plan to Share IPD: No